CLINICAL TRIAL: NCT01716793
Title: Risk Adapted Treatment for Primary AML in Adults up to the Age of 60 Years.
Brief Title: Risk-adapted Therapy for Adult Acute Myeloid Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-99
Record Dates: First submitted 2012-10-22; First posted 2012-10-30 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Primary AML; Risk-adapted treatment; Hematopoietic transplantation; CD34+ cell selection
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Risk-adapted postremission treatment (Other): Ara-C, autologous transplantation, Allogeneic HLA-identical sibling transplantation depending on risk factors (cytogenetics, courses to CR)and availability of an HLA-identical sibling, CD34+ selection.
  Interventions: Drug: Ara-C; Other: Autologous transplantation; Other: Allogeneic HLA-identical sibling transplantation; Other: CD34+ selection

INTERVENTIONS:
Drug: Ara-C — * Intermediate dose during induction phase to remission.
  * High-dose during consolidation phase in patients with favorable cytogenetics.
Other: Autologous transplantation — * In patients with normal karyotype and one cycle of chemotherapy to achieve complete remission.
  * In patients with other cytogenetics without HLA-Identical sibling.
Other: Allogeneic HLA-identical sibling transplantation — * Patients without favorable or normal karyotype(and one course to CR).
  * Patients with normal karyotype who need two cycles of chemotherapy to achieve CR, and other cytogenetics.
Other: CD34+ selection — In allotransplants, it is performed a CD34+ cell selection of peripheral blood stem cell transplantation.

SUMMARY:
In a protocol of treatment of AML used in 1994 for adults with AML up to the age of 50 years, the Spanish CETLAM group showed a complete remission rate 75 % using the combination of daunorubicin (60 mg/m2, 3 days) plus conventional dose cytarabine (100mg/m2/day in continuous infusion during 7 days) and etoposide (100mg/m2 IV/day 3 days). If idarubicin (10 mg/m2, 3 days) was administered instead of daunorubicin, the complete remission (CR) rate in adults up to 60 years was 75%. To improve the proportion of CRs and to decrease relapse rate appearing in 50% of patients, the phase II AML-99 trial includes intermediate dose-cytarabine during induction and risk-adapted post remission treatment based on the improvement in prognostic characterization of AML and the implementation of novel transplantation techniques.

DETAILED DESCRIPTION:
Induction chemotherapy: idarubicin (12mg/m2/day intravenous), intermediate-dose cytarabine (500mg/m2/12h, intravenous) and etoposide (100mg/m2/day, intravenous) in 3+7+3 schedule. This induction therapy is repeated if complete remission (CR) is not achieved after the first course of treatment.

Consolidation therapy: mitoxantrone (12mg/m2/day, intravenous, days 4, 5 and 6) and intermediate-dose cytarabine (500mg/m2/12h from day 1 to 6).

Risk-stratification according to cytogenetics, courses to CR and availability of an HLA-identical sibling:

* Patients in the favorable cytogenetics group [t(8;21), inv(16) or t(16;16)] are treated with high-dose cytarabine (3g/m2/12h, intravenous, days 1, 3 and 5).
* Patients in intermediate cytogenetics group (normal karyotype and a single course to achieve the CR) receive an autologous peripheral blood stem cell (PBSC) transplant, regardless of having an HLA-identical sibling.
* The remaining patients are considered in the high-risk group and are treated with autologous or allogeneic PBSC transplantation depending on the availability of a sibling donor. In allotransplants, CD34+ cell selection of hematopoietic cells is performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML, classified by FAB criteria
* Age not superior to 60 years
* Verbal informed consent for the chemotherapy and written for the mobilization and stem cell transplantation

Exclusion Criteria:

* Patients treated previously for its AML with other chemotherapy different from hydroxyurea
* Acute promyelocytic leukemia (M3)
* Chronic myeloid leukemia in blastic crisis
* Leukemias appearing after other myeloproliferative processes
* Leukemias surviving after myelodysplastic syndromes with more than 6 months of evolution
* Presence of other neoplastic disease in activity
* Secondary AML which had appeared after cured malignancies (for instance Hodgkin disease) and those who are still exposed to alkylant agents or radiation
* Renal and hepatic abnormal function with creatinine values and/or bilirubin two times higher than the normal threshold, except when this alteration could be attributed to the leukemia
* Patients with a fraction of ejection very low (inferior to 40%), symptomatic cardiac insufficiency or both
* Patients with a grave concomitant neurological or psychiatric disease
* Positivity of HIV (donor and/or receptor)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 1998-09; Primary Completion 1998-09 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Complete remission rate. | 2 months.
  Analyze the efficacy and toxicity of IDICE (idarubicin, intermediate doses of ara-C and etoposide) to achieve complete remission.
Disease free survival. | 4 years.
  Analyze the disease free survival (DFS)of patients in remission, with a therapeutic strategy adjusted to the prognostic factors.

SECONDARY OUTCOMES:
Evaluations of minimal residual disease (MRD) by flow cytometry during and after treatment. | 4 years.
  Study of the immunophenotypic characteristics of the leukemic population at diagnosis and evaluation of MRD during different treatment phases and follow-up.
Feasibility to mobilize and collect autologous PBSC after consolidation phase. | 6 months.
  Evaluation of mobilization failures.
Evaluations of the CD34+ cell selection procedure and allogeneic peripheral blood stem cell (PBSC)transplantation outcome. | 4 years.
  CD34+ cell selection from PBSC of HLA-identical siblings. Conditioning regimen. Infusion and post-transplant follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sierra, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Salut Brunet, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (19):
- Spain (19):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Centro Medico Teknon, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Jordi Esteve, Barcelona, Barcelona
  - ICO Hospital Universitari de Bellvitge, L'Hospitalet Del Llobregat, Barcelona
  - Hospital A Coruña, A Coruña, Coruña
  - Hopital Universitari de Girona Dr. Josep Trueta, Girona, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida, Lleida
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Joan Bargay, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Murcia, Murcia, Murcia
  - Hospital Universitari Joan XXIII, Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Mutua de Terrassa, Terrassa, Terrassa
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid, Valladolid